CLINICAL TRIAL: NCT07147933
Title: Physical Therapy Protocol for Crouch Gait Associated to the Anterior Pelvic Tilt and Soleus Muscle Weakness in CP Patient
Brief Title: Effect of Treatment on Cerebral Palsy Patient With Crouch Gait Associated With Anterior Pelvic Tilt and Soleus Muscle Weakness"Marouf Syndrome", and Muscle Assesment by Using EMG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Philadelphia University, Jordan (Other)
Responsible Party: Principal Investigator, Ahmed Yasser Mostafa Marouf, physical therapist (BSc PT), Philadelphia University, Jordan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2/5/2024-2025
Record Dates: First submitted 2025-08-22; First posted 2025-08-29 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy (CP); Diaplegia; Muscle Weakness | Patient; Anterior Pelvic Tilt; Crouch Gait
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled trial designed using a parallel assignment model. Participants will be randomly divided into two groups. One group will receive the physical therapy intervention being studied, while the other group will receive tradtional physical therapy protocol. The aim is to compare the effects of the intervention by measuring muscle activity using surface electromyography (sEMG) before and after the treatment.
Who Masked: Outcomes Assessor
Masking Description: (single blind) the Outcomes Assessor who was unaware to the approach of treatment that would be executed to the children into two groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): A targeted physical therapy program including correction of anterior pelvic tilt, strengthening of the soleus, core strengthening, stretching of the hamstrings, and strengthening of the quadriceps. The program will be delivered 3 times per week for 8 weeks under therapist supervision.
  Interventions: Other: phusical therapy program; Other: physical therapy program
- Arm B (Active Comparator): physical therapy program including stretching of the hamstrings and strengthening of the quadriceps only. The program will be delivered 3 times per week for 8 weeks under therapist supervision
  Interventions: Other: phusical therapy program; Other: physical therapy program

INTERVENTIONS:
Other: phusical therapy program — physical therapy program including stretching of the hamstrings and strengthening of the quadriceps only. The program will be delivered 3 times per week for 8 weeks under therapist supervisio
Other: physical therapy program — A targeted physical therapy program including correction of anterior pelvic tilt, strengthening of the soleus, core strengthening, stretching of the hamstrings, and strengthening of the quadriceps. The program will be delivered 3 times per week for 8 weeks under therapist supervision.

SUMMARY:
Children with cerebral palsy (CP) often develop gait abnormalities, with crouch gait being a common and challenging issue that affects their posture and daily function. Numerous studies indicate that crouch gait is primarily caused by hamstring tightness and quadriceps weakness. Traditional treatment approaches focus on hamstring stretching and quadriceps strengthening exercises to improve gait patterns. highlight the importance of strengthening muscles like the quadriceps and stretching tight muscles such as the hamstrings in improving gait abnormalities source.

Despite these common treatments, results often fall short of achieving full correction of crouch gait. Therefore, I propose a novel approach to treating abnormal gait in children with CP by targeting the anterior pelvic tilt and strengthening the soleus muscle. This approach aims to address biomechanical factors that are not typically considered in traditional treatments, potentially leading to better functional outcomes

we use Surface EMG to record activity of key muscle (soleus) during Seated Calf Raises exercise Muscle activity will be recorded before and after a series of physical therapy sessions focused on pelvic alignment and soleus strengthening.

EMG Data Analysis: Root Mean Square (RMS), timing of activation, and amplitude changes will be assessed.

ELIGIBILITY:
Inclusion Criteria:

patient with cp have a crouch gait. ages from 4 to 10 years . have a anterior pelvic tilt . muscle weakness (Soleus) on EMG.

* BMI from 18.5 to 21..
* didn't submit to Selective Dorsal Rhizotomy surgery.

Exclusion Criteria:

have a posterior pelvic tilt.

-above 10 or below 4 years. not able to walk. . submitted to SDR surgery. BMI above 21 or below 18.5.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-03-02 (Estimated); Study Completion 2026-03-02 (Estimated)

PRIMARY OUTCOMES:
EMG and we calculate RMS for soleus muscle | the primary outcome measures by using EMG before treatment paln and after 8 weeks

SECONDARY OUTCOMES:
step length | before treatment plan and after 8 weeks
step wedth | before treatment plan and after 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Yasser Mostafa Marouf, bachelor's physical thrapy, Principal Investigator — Bachelor's of Physical Therapy, Faculty of Allied Medical Sciences, Philadelphia University, Amman; Mayar Mostafa Rady Abdelmogaly, bachelor's physical thrapy, Study Director — Mayar Mostafa Rady Abdelmogaly Bachelor's of physical therapy, Galala university
Locations (1):
- Queen Rania AL Abdullah hospital for children, Amman, Jordan

IPD SHARING:
Plan to Share IPD: Undecided